CLINICAL TRIAL: NCT07210489
Title: Therapeutic Benefits of a Motor Imaging Protocol After Anterior Cruciate Ligament Reconstruction Surgery: Study of Lower Limb Symmetry During Various Functional Tests
Brief Title: Therapeutic Benefits of a Motor Imaging Protocol Following Anterior Cruciate Ligament Reconstruction Surgery
Acronym: IMAGERIEMOTR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025-A01415-44
Record Dates: First submitted 2025-09-19; First posted 2025-10-07 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Anterior Cruciate Ligament Tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Prospective, comparative, randomized, controlled, single-blind (patient), single-center study
Who Masked: Participant
Masking Description: single-blind (patient)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor imagery program (Experimental): Patients will receive rehabilitation sessions from a physical therapist in accordance with standard practice and will be asked to complete a 3-week motor imagery program starting 3 months after anterior cruciate ligament surgery.
  Interventions: Procedure: Reconstructive surgery after anterior cruciate ligament rupture; Other: sessions from a physical therapist
- Cognitive (non-motor) task program (Active Comparator): Patients will receive rehabilitation sessions from a physical therapist in accordance with standard practice and will be asked to complete a 3-week cognitive (non-motor) task program starting 3 months after anterior cruciate ligament surgery.
  Interventions: Procedure: Reconstructive surgery after anterior cruciate ligament rupture; Other: sessions from a physical therapist

INTERVENTIONS:
Procedure: Reconstructive surgery after anterior cruciate ligament rupture — surgical technique for repairing the cruciate ligament
Other: sessions from a physical therapist — sessions from a physical therapist in accordance with standard practice

SUMMARY:
The purpose of this study is to compare changes in lower limb symmetry during functional and strength tests, before and after the motor imagery program, in patients who received the 3-week motor imagery program starting 3 months post-surgery versus patients who did not receive the motor imagery program.

DETAILED DESCRIPTION:
This is a prospective, comparative, randomized, controlled, single-blind (patient), single-center study evaluating the effects of a motor imagery program in parallel with rehabilitation sessions in patients who have had an anterior cruciate ligament rupture.

The study population is composed of adult patients who underwent reconstructive surgery after anterior cruciate ligament rupture, followed up at the Clinique de la Sauvegarde in Lyon for post-operative functional and strength testing of the anterior cruciate ligament.

Patients included in the study will be randomized into two study arms (experimental arm and control arm).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 45;
* Individuals who have undergone anterior cruciate ligament reconstruction for the first time on the operated leg;
* All types of surgery (harvesting of the new gracilis or patellar tendon) within 3 months prior to inclusion;
* Patients able to understand and read French;
* Affiliation with a social insurance plan;
* Signed informed consent.

Exclusion Criteria:

* Recurrence or rupture of the contralateral anterior cruciate ligament;
* Osteotomy;
* Cognitive disorders observed by the investigator;
* Vestibular disorders known to the patient or observed by the investigator;
* Post-surgical complications (infection, early graft rupture);
* Patient participating in another interventional clinical trial, or in a period of exclusion from another interventional study;
* Patient under guardianship or conservatorship;
* Pregnant or breastfeeding women.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Evolution of limb symmetry | between 3 and 4.5 months
  Evolution of limb symmetry assessed by the Limb Symmetry Index in %
Isometric quadriceps strength | between 3 and 4.5 months
  Isometric quadriceps strength using a Micro Fet handheld dynamometer (in Newtons)
Isometric hamstring strength | between 3 and 4.5 months
  Isometric hamstring strength measured using a Micro Fet handheld dynamometer (in Newtons)
Average concentric strength | between 3 and 4.5 months
  Average concentric strength during a counter-movement jump measured using a force platform (in Newtons)
Average strength | between 3 and 4.5 months
  Average strength during a squat measured using a force platform (in Newtons)
Quadriceps activation measured | between 3 and 4.5 months
  Quadriceps activation measured using electromyography

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique de la Sauvegarde, Lyon, France